CLINICAL TRIAL: NCT00403611
Title: Evaluation of Praziquantel Dosage for Treatment of Schistosomiasis in Highly Endemic Areas of Northeastern Brazil
Brief Title: Evaluation of Praziquantel Dosage for Treatment of Schistosomiasis in Brazil
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: World Health Organization (Other); Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Otavio Sarmiento Pieri, Senior Researcher, Oswaldo Cruz Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A20764
Record Dates: First submitted 2006-11-24; First posted 2006-11-27 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Schistosomiasis Mansoni
MeSH Terms: conditions — Schistosomiasis mansoni | interventions — Praziquantel

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Praziquantel 40mg/kg (Active Comparator): Praziquantel (Distocide) 40mg/kg single oral dose
  Interventions: Drug: Praziquantel 40 mg/kg
- Praziquantel 60mg/kg (Experimental): Praziquantel (Distocide) 60mg/kg single oral dose
  Interventions: Drug: Praziquantel 60 mg/kg

INTERVENTIONS:
Drug: Praziquantel 60 mg/kg — Praziquantel (Distocide) 60 mg/kg single oral dose
  Other Names: Distocide
  Arms: Praziquantel 60mg/kg
Drug: Praziquantel 40 mg/kg — Praziquantel (Distocide) 40 mg/kg single oral dose
  Other Names: Distocide
  Arms: Praziquantel 40mg/kg

SUMMARY:
The primary objective of this project is to evaluate the efficacy and safety of praziquantel 60 mg/kg in the treatment of schistosomiasis, as compared to the standard 40 mg/kg therapy in a representative community from a highly endemic area of schistosomiasis in Northeastern Brazil. Cure rates, reduction in egg counts and proportions of reported side-effects in children at the 10-19 y age-range with at least 100 eggs per gram of faeces will be compared between regimens, aiming to evaluate the superiority of 60 mg/kg over the 40mg/kg dose currently recommended by the WHO. Reinfection rates will also be evaluated aiming to improve transmission control within the local health system, including re-treatment combined with auxiliary control measures. Features related to the clinical, nutritional and immunological status of the patients prior to treatment will also be investigated in association with the outcome of praziquantel treatment.

DETAILED DESCRIPTION:
This is a double blind, randomized, PZQ 40mg/Kg- controlled clinical trial. Subjects 10-19 years old living in communities of the Northeast of Brazil will be identified and invited to participate in this study.

Well trained field health agents will first make a sketch map of the village (depicting the location of houses, main water courses, snail habitats and water-contact sites) and apply a household questionnaire to obtain personal data from residents to identify the individuals in the 10-19 years age range, as well as to record sanitary standards of the houses and water-contact reported behaviour as described by Pieri et al. (1998, Mem. Inst. Oswaldo Cruz, 93, Suppl 1: 259-264).

Meetings with the Caricé Community Association will be held in order to explain to the inhabitants the purpose, the objectives of the study, and how the study will be conducted.

Thereafter, all residents between 10 and 19 yrs of age will be interviewed at their homes regarding the fulfilment of the inclusion/exclusion criteria. Those who fulfil the criteria and agree to participate in the screening phase of the trial (signed Screening Informed Consent) will be given stool vials and asked to provide stool samples (two samples within 5-day intervals) that will be collected at their homes in the following days, stored in heat-proof containers and taken to the premises of the Service of Reference for Schistosomiasis Diagnosis of the CPqAM to be promptly prepared for examination by the Kato-Katz method (Katz et al, 1972, Rev. Inst. Med. Trop. Sao Paulo, 14: 397-400) aiming to identify positive cases and estimate individual egg load. Females on childbearing age will also be asked to provide a urine sample for pregnancy test. Pregnant women will only be treated with Praziquantel after weaning, as currently recommended by Funasa, and will be excluded from the trial. The 2 stool samples provided by each individual will be analysed for S. mansoni infection. Two slides will be prepared from each stool sample, and the mean value of the 4 slides (as measured by number of eggs/g of stool) will be calculated. Only those harbouring at least 100 epg who are able and willing to follow-up will be invited to participate in the study. At this stage, individuals with positive diagnosis for S. mansoni and that for any reason were excluded from the study will receive standard treatment for schistosomiasis.

In the enrolment visit the subjects eligible for the study, will be examined by the physician and interviewed to assess inclusion/exclusion criteria. Those who fulfill all criteria will be invited to participate in the trial and will go through the Informed Consent Form procedure (see details in section 6.14). For those who accept to participate and provide a written Informed Consent: weight and height will be measured, a 5ml venous blood sample will be collected and an abdominal ultra-sound exam will be performed. After all these procedures, the patient will be assigned to the treatment.

Subjects will be randomly allocated to either Group A (single 40 mg/kg oral dose) or Group B (single 60 mg/kg oral dose), as described in sections 6.4.3 and 6.4.4. Praziquantel tablets will be provided by TDR. During four hours after treatment the subjects will be observed for safety assessment, and one day and 21 days after treatment they will be interviewed about the following symptoms related to praziquantel side-effects: abdominal pain, diarrhea, vomiting, nausea, drowsiness, general malaise, edema, skin rash, urticaria, myalgia, heartburn, fever, dizziness and headache (Guisse et al, 1997, Am. J. Trop. Med. Hyg., 56: 511-514, 1997). The follow-up visits to assess efficacy and morbidity will be at 21 days, six months and 12 months after treatment, when the subjects will be surveyed by the Kato-Katz method (two stool samples within five-day interval, two slides each). Weight and height will be measured at 6 and 12 months follow-up. Ultrasound will be repeated at 6 and 12 months follow-up visits for the participants who presented periportal fibrosis or liver/spleen enlargement in the baseline (D0) exam.

ELIGIBILITY:
Inclusion Criteria:

* Persons with 10-19 years of age harbouring at least 100 epg who are able and willing to follow-up and provide a written informed consent will participate in the study

Exclusion Criteria:

* Pregnancy or lactation
* Acute or chronic severe diseases including hepato-splenic schistosomiasis
* Use of praziquantel in the last 30 days
* Known hypersensitivity associated with praziquantel
* Current use of other medication that may affect the results of the present trial, such as antibiotics and corticosteroids, and any medical condition that on the judgement of the physician makes subject participation impossible.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 196 (Actual)
Dates: Start 2006-03; Primary Completion 2007-10 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Cure rate and egg reduction rate at twenty-one days after treatment | 21 days

SECONDARY OUTCOMES:
Occurrence of the following symptoms following praziquantel administration: abdominal pain, diarrhea, vomiting, nausea, drowsiness, general malaise, edema, skin rash, urticaria, myalgia, heartburn, fever, dizziness and headache. | 21 days
Weight (Kg) and height (m) measured at Day 0, 6 months and 12 months follow-up visits. | 12 months
Presence/absence of periportal fibrosis and liver or spleen enlargement at Day 0, 6 months and 12 months follow-up visits. | 12 months
Factors associated with cure/failure at Day 21 evaluation: | 21 days
Haematological: Haemoglobin/ Hematocrit, leukocytes count, lymphocytes and eosinophiles count. | 0 days
Biochemistry: liver function will be evaluated by serum bilirubin, alkaline phosphatase, aspartate aminotransferase, and alamin aminotransferase levels. | 0 days
Immunological: Titles of anti-SEA and anti-SWAB antibodies. | 0 days
Reinfection rate and Egg reduction rate at six and twelve months after treatment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Otavio S Pieri, PhD, Principal Investigator — Fundação Oswaldo Cruz; Ana Lucia C Domingues, MD, Principal Investigator — Universidade Federal de Pernambuco